CLINICAL TRIAL: NCT00508755
Title: Feasibility and Practice Characteristics of FNS and Gait Robot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B4036-I
Record Dates: First submitted 2007-07-27; First posted 2007-07-30 (Estimated); Results first posted 2014-04-02 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Stroke
Keywords: cerebrovascular accident; electrical stimulation; gait training; motor learning
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): stroke
  Interventions: Device: Gait Robot; Device: Functional Neuromuscular stimulation with intramuscular electrodes

INTERVENTIONS:
Device: Gait Robot — gait training with the use of a gait robot
Device: Functional Neuromuscular stimulation with intramuscular electrodes — gait training with use of functional electrical stimulation

SUMMARY:
Conventional therapies do not restore normal gait for many stroke survivors. The long-term goal of this work is to restore volitional lower limb motor control and gait following stroke. In our prior work, we demonstrated that it was feasible to provide a clinically operated, combined treatment of body weight supported treadmill training alone (BWSTT) + functional neuromuscular stimulation (FNS) using intramuscular (IM) electrodes (FNS-IM).

Specific Aims and Hypothesis The purpose or Specific Aim of the study is to test the feasibility and gait training potential of combining the Lokomat and FNS-IM for stroke survivors. Given the feasibility of our clinically operated combination of BWSTT + FNS-IM, we propose to test the feasibility of the combination of Lokomat + FNS-IM.

Hypothesis I. It is feasible to utilize a clinically operated combination of Lokomat + functional neuromuscular stimulation (FNS) with intramuscular (IM) electrodes (FNS-IM).

Treatment Procedures. The subjects will be treated for three months, four sessions/week (for a total of 48 treatment visits). A given session will be 1 hrs, with the time divided into thirds as follows: 1) hr coordination exercise; 2) hr over ground gait training; and 3) hr Lokomat gait training. FNS-IM will be used in all three aspects of the protocol, unless the subject is capable of volitionally executing a given movement or gait component. Population. The subjects will be chronic stroke survivors (>6 months after the stroke).

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 6 months after stroke
* 21 years or older
* Ability to follow 2 step commands
* Inability to move leg normally

Exclusion Criteria:

* Pacemaker
* Progressive medical condition (i.e. Parkinsons Disease)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2005-08; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janis Daly, PhD MS, Principal Investigator — VA Medical Center-Cleveland
Locations (1):
- VA Medical Center, Cleveland, Cleveland, Ohio, United States

REFERENCES:
- [Result] McCabe JP, Dohring ME, Marsolais EB, Rogers J, Burdsall R, Roenigk K, Pundik S, Daly JJ. Feasibility of combining gait robot and multichannel functional electrical stimulation with intramuscular electrodes. J Rehabil Res Dev. 2008;45(7):997-1006. doi: 10.1682/jrrd.2007.08.0124. PMID 19165689
- [Result] Dohring ME, Daly JJ. Automatic synchronization of functional electrical stimulation and robotic assisted treadmill training. IEEE Trans Neural Syst Rehabil Eng. 2008 Jun;16(3):310-3. doi: 10.1109/TNSRE.2008.920081. PMID 18586610

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited through use of advertisement and by word of mouth to enter this feasibility study.
Groups:
- Gait Training After Stroke: Subjects with chronic stroke (.5-1.5 years post stroke) received gait training with the use of functional neuromuscular stimulation with intramuscular electrodes and gait robot.
Period: Overall Study
Arm/Group | Gait Training After Stroke
Started | 6
Completed | 5
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: This was a feasibility study of six subjects. Sample size was constrained by funding limit.
Arm/Group | Gait Training After Stroke
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Observational Gait Components: Observational Comparison of Gait Components for: Gait Robot-alone Condition, FES-alone Condition, and Combined Gait Robot and FES.
Description: Observational Gait components during stance and swing phase, for pelvis, hip, knee, and ankle for each of the six participants was observed during the following conditions: Gait Robot-alone, FES-alone, and combined Gait Robot and FES.
Time Frame: visit 48, following treatment
Population: The sample size for this feasibility study was n=6, constrained by funding limit.
Measure: Number; unit: participants
Groups:
- Gait Robot-alone Training: The 6 study subjects with chronic stroke ambulated in the Gait Robot, and observational gait analysis was performed.
- FES-Alone: The 6 study subjects with chronic stroke ambulated with FES, and observational gait analysis was performed.
- Combined Gait Robot and FES: The 6 study subjects with chronic stroke ambulated with combination Gait Robot and FES, and observational gait analysis was performed.
Arm/Group | Gait Robot-alone Training | FES-Alone | Combined Gait Robot and FES
Number analyzed (Participants) | 6 | 6 | 6
participants
  allowed for lateral weight shift | 0 | 6 | 6
  allowed for knee control-stance phase | 6 | 6 | 6
  allowed for ankle movement in sagittal plane | 6 | 6 | 6

ADVERSE EVENTS:
Groups:
- Gait Training After Stroke: subjects with Chronic stroke (.5-1.5 years post stroke)received gait training with the use of functional neuromuscular stimulation with intramuscular electrodes and Gait Robot.
Arm/Group | Gait Training After Stroke
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
This was a feasibility study to determine the possibility of combining two technologies. Further study of the combined treatment is needed to determine whether the feasible combined treatment is more effective than other methods.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes